CLINICAL TRIAL: NCT00377312
Title: Determining the Maximal Safe Dose of a Continuous Infusion of Parathyroid Hormone(1-34): Effects on Bone Formation
Brief Title: 7 Day Continuous Parathyroid Hormone IV Infusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor of Medicne, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 0606127; R01DK073039 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis; Bone Diseases, Endocrine; Hyperparathyroidism
Keywords: Endocrine System Diseases; MusculoSkeletal System Disease; Hormone; Physiologic Properties
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Endocrine; Hyperparathyroidism; Endocrine System Diseases; Musculoskeletal Diseases | interventions — Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Parathyroid Hormone (PTH) (1-34) 2 picomols/kg/hr for one week.
  Interventions: Drug: Parathyroid Hormone (1-34)
- Group 2 (Experimental): Parathyroid Hormone (PTH) (1-34)4 picomols/kg/hr for one week.
  Interventions: Drug: Parathyroid Hormone (1-34)

INTERVENTIONS:
Drug: Parathyroid Hormone (1-34) — PTH(1-34) IV given over a one week period
  Other Names: IND 60,979

SUMMARY:
Study consists of an eight day inpatient visit on the General Clinical Research Center. The investigators' specific aims are to:

1. To define the maximum safe dose of a seven day continuous administration of parathyroid hormone [PTH(1-34)] in healthy human volunteers.
2. To estimate the effect of a seven day continuous administration of parathyroid Hormone (PTH) in escalating doses on vitamin D metabolism, markers of bone turnover and fractional excretion of urine.

DETAILED DESCRIPTION:
This study will expand upon earlier infusions studies that demonstrated: 1) There is a dose-related increase in 1,25 (OH)2 vitamin D in response to PTHrP and PTH over multiple days. 2) There is a markedly attenuated vitamin D response to PTHrP compared to PTH, particularly during the second 24 hours. 3) The increase in 1,25 (OH)2 vitamin D is almost certainly responsible for the greater calcemic effect of PTH compared to PTHrP. 4) PTHrP is obviously a weaker agonist of 1,25 (OH)2 vitamin D but does not result in its suppression as is seen in Humoral Hypercalcemia of Malignancy (HHM). Thus, the suppression of 1,25 (OH)2 vitamin D seen in HHM remained unexplained. In addition to assessing the effects of an infusion of PTHrP and PTH on calcium handling and 1,25(OH)2 vitamin D, we also measured their effects on markers of bone turnover. Given the clinical observations seen in Hyperparathyroidism (HPT) and HHM, we anticipated that PTH would stimulate both bone resorption and formation, while PTHrP would stimulate bone resorption but inhibit formation. However, we observed that infusions of PTHrP and PTH resulted in an equivalent, rapid increase in bone resorption as measured by N-telopeptide (NTx) and C-telopeptide (CTx), as well as a progressive decline in bone formation. There was no difference between PTH and PTHrP. We assumed that formation would ultimately increase with additional time, as seen in HPT, and therefore examined an additional group of subjects infused with PTHrP for 96 hours. However, N-terminal propeptide of type 1 procollagen (P1NP) continued to decline even further as is seen in HHM in contrast to HPT. We have not yet studied longer infusions of PTH.

One of the reasons for doing this pilot study is to determine the optimal dosing of PTH over a week period of time. Intravenous PTH has never been infused into human beings for prolonged periods of time. The investigators question whether a prolonged continuous intravenous infusion of PTH will lead to a sustained and progressive suppression of bone formation as occurs in HHM or an increase in bone formation as occurs in HPT. They also want to assess the direct influence of long-term continuous PTH infusions on plasma 1,25 (OH)2 vitamin D regulation in healthy human volunteers. We have shown in our previous studies that doses of 8 picomoles (pmol)/kg/hr PTH given over 48 hours result in sustained mild serum hypercalcemia, with serum calcium seeming to plateau in the range of 11 - 11.5 mg/dL after 48 hours. A dose of 8 picomoles (pmol)/kg/hr has also been shown to cause desirable effects on serum 1,25(OH)2 vitamin D and markers of bone turnover, and may therefore be the "ideal" dose. However, we do not know whether serum calcium will plateau after an infusion of 48 hours with escalating doses or whether it will continue to increase over seven days.

To determine what will happen with a prolonged infusion, we plan to start with doses lower than 8 picomoles (pmol)/kg/hr, and then gradually increase the dose of PTH in successive groups of subjects. In the event of a significant adverse effect, immediate action will be taken to reverse it. Protocols will be in place to follow in the event of expected adverse events such as hypotension, nausea, and muscle cramping. Severe sudden side effects are not anticipated; however, mild easily reversible side effects are to be expected as an outcome in order to determine the optimal dose of PTH. This study has been approved by the NIH and the Data Safety Monitoring Board (DSMB).

Seventy five normal healthy men and women will be screened for an eight day in-patient admission to the General Clinical Research Center (GCRC). Thirty evaluable research participants will receive a seven day infusion of a predetermined dose of PTH. Vitals signs, blood pressure, blood and urine lab results will be monitored frequently as per the study flow sheet. The starting dose of PTH, 2 picomoles (pmol)/kg, will be given to three normal healthy subjects. The dose will be escalated in increments with successive groups of three subjects each, until early adverse effects (mild hypercalcemia, postural hypotension, tachycardia) are seen. This dose will then be used in future studies. The investigators with this study are trying to discover if a prolonged continuous intravenous infusion of PTH will lead to a sustained and progressive suppression of bone formation as occurs in HHM or an increase in bone formation as occurs in HPT.

Subject Population will consist of healthy young adults, ages 24-35 years, as in our other safety and physiologic studies. It is anticipated that we will need to screen 75 subjects in order to obtain 30 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian, Hispanic or Asian subjects
* Males and Females
* Non-smoker
* Ages 24 - 35 years old
* Subjects will be recruited either from the employee pool of the University of Pittsburgh or the University of Pittsburgh Medical Center (UPMC), or the general population living in the vicinity.
* Participation in this study by an employee or a potential employee at the University of Pittsburgh or UPMC has no effect on their employment or potential employment.
* Participants in the study will be required to discontinue all vitamins and health food supplements two weeks prior to the study.

Exclusion Criteria:

* Cardiac, hypertensive, vascular, renal (serum creatinine of >1.5), pulmonary, endocrine, musculoskeletal, hepatic, hematologic or malignant or rheumatologic disease
* Body Mass Index (BMI) > 30,
* Anemia (hematocrit less than 36% in women, less than 40% in men),
* Pregnancy (all women will have a urine pregnancy test performed immediately before starting the study and must not be pregnant)
* Significant alcohol or drug abuse or
* Baseline hypotension (systolic blood pressure less than 90 mm/Hg).
* Subjects will be excluded for abnormal levels of any of the screening labs including: ionized and total serum calcium, phosphorus, creatinine, albumin, 25-hydroxyvitamin D, and PTH. Pregnancy
* Subjects taking any chronic medications except oral contraceptives and stable doses of thyroid hormone, or those who have received any investigational drug in past 90 days will be excluded from the study.
* Subjects may not participate in this study more than once.
* Any subject who has previously received PTH or PTHrP, a related peptide, may not participate in this study.

Minority Inclusion/Exclusion Statement: We will not include African-Americans because this group has been demonstrated by a number of investigators to display resistance to PTH, and may create wider statistical variation and a need for larger numbers of study subjects per group.

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara J. Horwitz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horwitz MJ, Tedesco MB, Gundberg C, Garcia-Ocana A, Stewart AF. Short-term, high-dose parathyroid hormone-related protein as a skeletal anabolic agent for the treatment of postmenopausal osteoporosis. J Clin Endocrinol Metab. 2003 Feb;88(2):569-75. doi: 10.1210/jc.2002-021122. PMID 12574182
- [Background] Syed MA, Horwitz MJ, Tedesco MB, Garcia-Ocana A, Wisniewski SR, Stewart AF. Parathyroid hormone-related protein-(1--36) stimulates renal tubular calcium reabsorption in normal human volunteers: implications for the pathogenesis of humoral hypercalcemia of malignancy. J Clin Endocrinol Metab. 2001 Apr;86(4):1525-31. doi: 10.1210/jcem.86.4.7406. PMID 11297578
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Everhart-Caye M, Inzucchi SE, Guinness-Henry J, Mitnick MA, Stewart AF. Parathyroid hormone (PTH)-related protein(1-36) is equipotent to PTH(1-34) in humans. J Clin Endocrinol Metab. 1996 Jan;81(1):199-208. doi: 10.1210/jcem.81.1.8550752.
- [Background] Henry JG, Mitnick M, Dann PR, Stewart AF. Parathyroid hormone-related protein-(1-36) is biologically active when administered subcutaneously to humans. J Clin Endocrinol Metab. 1997 Mar;82(3):900-6. doi: 10.1210/jcem.82.3.3811. PMID 9062504
- [Background] Plotkin H, Gundberg C, Mitnick M, Stewart AF. Dissociation of bone formation from resorption during 2-week treatment with human parathyroid hormone-related peptide-(1-36) in humans: potential as an anabolic therapy for osteoporosis. J Clin Endocrinol Metab. 1998 Aug;83(8):2786-91. doi: 10.1210/jcem.83.8.5047. PMID 9709948
- [Background] Stewart AF, Cain RL, Burr DB, Jacob D, Turner CH, Hock JM. Six-month daily administration of parathyroid hormone and parathyroid hormone-related protein peptides to adult ovariectomized rats markedly enhances bone mass and biomechanical properties: a comparison of human parathyroid hormone 1-34, parathyroid hormone-related protein 1-36, and SDZ-parathyroid hormone 893. J Bone Miner Res. 2000 Aug;15(8):1517-25. doi: 10.1359/jbmr.2000.15.8.1517. PMID 10934650
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Garcia-Ocana A, Bisello A, Hollis BW, Gundberg C, Stewart AF. Safety and tolerability of subcutaneous PTHrP(1-36) in healthy human volunteers: a dose escalation study. Osteoporos Int. 2006 Feb;17(2):225-30. doi: 10.1007/s00198-005-1976-3. Epub 2005 Sep 7. PMID 16151606
- [Background] Juppner H, Abou-Samra AB, Freeman M, Kong XF, Schipani E, Richards J, Kolakowski LF Jr, Hock J, Potts JT Jr, Kronenberg HM, et al. A G protein-linked receptor for parathyroid hormone and parathyroid hormone-related peptide. Science. 1991 Nov 15;254(5034):1024-6. doi: 10.1126/science.1658941.
- [Background] Orloff JJ, Wu TL, Heath HW, Brady TG, Brines ML, Stewart AF. Characterization of canine renal receptors for the parathyroid hormone-like protein associated with humoral hypercalcemia of malignancy. J Biol Chem. 1989 Apr 15;264(11):6097-103. PMID 2539369
- [Background] Orloff JJ, Ribaudo AE, McKee RL, Rosenblatt M, Stewart AF. A pharmacological comparison of parathyroid hormone receptors in human bone and kidney. Endocrinology. 1992 Oct;131(4):1603-11. doi: 10.1210/endo.131.4.1327716.
- [Background] Samuels MH, Veldhuis J, Cawley C, Urban RJ, Luther M, Bauer R, Mundy G. Pulsatile secretion of parathyroid hormone in normal young subjects: assessment by deconvolution analysis. J Clin Endocrinol Metab. 1993 Aug;77(2):399-403. doi: 10.1210/jcem.77.2.8345044.
- [Background] Prank K, Nowlan SJ, Harms HM, Kloppstech M, Brabant G, Hesch RD, Sejnowski TJ. Time series prediction of plasma hormone concentration. Evidence for differences in predictability of parathyroid hormone secretion between osteoporotic patients and normal controls. J Clin Invest. 1995 Jun;95(6):2910-9. doi: 10.1172/JCI117998. PMID 7769133
- [Background] Schmitt CP, Obry J, Feneberg R, Veldhuis JD, Mehls O, Ritz E, Schaefer F. Beta1-adrenergic blockade augments pulsatile PTH secretion in humans. J Am Soc Nephrol. 2003 Dec;14(12):3245-50. doi: 10.1097/01.asn.0000101240.47747.7f. PMID 14638923
- [Background] Chapotot F, Gronfier C, Spiegel K, Luthringer R, Brandenberger G. Relationships between intact parathyroid hormone 24-hour profiles, sleep-wake cycle, and sleep electroencephalographic activity in man. J Clin Endocrinol Metab. 1996 Oct;81(10):3759-65. doi: 10.1210/jcem.81.10.8855835.
- [Background] Harms HM, Schlinke E, Neubauer O, Kayser C, Wustermann PR, Horn R, Kulpmann WR, von zur Muhlen A, Hesch RD. Pulse amplitude and frequency modulation of parathyroid hormone in primary hyperparathyroidism. J Clin Endocrinol Metab. 1994 Jan;78(1):53-7. doi: 10.1210/jcem.78.1.8288713.
- [Background] Ledger GA, Burritt MF, Kao PC, O'Fallon WM, Riggs BL, Khosla S. Role of parathyroid hormone in mediating nocturnal and age-related increases in bone resorption. J Clin Endocrinol Metab. 1995 Nov;80(11):3304-10. doi: 10.1210/jcem.80.11.7593443.
- [Background] el-Hajj Fuleihan G, Klerman EB, Brown EN, Choe Y, Brown EM, Czeisler CA. The parathyroid hormone circadian rhythm is truly endogenous--a general clinical research center study. J Clin Endocrinol Metab. 1997 Jan;82(1):281-6. doi: 10.1210/jcem.82.1.3683. PMID 8989274
- [Background] Plawner LL, Philbrick WM, Burtis WJ, Broadus AE, Stewart AF. Cell type-specific secretion of parathyroid hormone-related protein via the regulated versus the constitutive secretory pathway. J Biol Chem. 1995 Jun 9;270(23):14078-84. doi: 10.1074/jbc.270.23.14078. PMID 7775469
- [Background] Fraher LJ, Hodsman AB, Jonas K, Saunders D, Rose CI, Henderson JE, Hendy GN, Goltzman D. A comparison of the in vivo biochemical responses to exogenous parathyroid hormone-(1-34) [PTH-(1-34)] and PTH-related peptide-(1-34) in man. J Clin Endocrinol Metab. 1992 Aug;75(2):417-23. doi: 10.1210/jcem.75.2.1322424.
- [Background] Burtis WJ, Wu T, Bunch C, Wysolmerski JJ, Insogna KL, Weir EC, Broadus AE, Stewart AF. Identification of a novel 17,000-dalton parathyroid hormone-like adenylate cyclase-stimulating protein from a tumor associated with humoral hypercalcemia of malignancy. J Biol Chem. 1987 May 25;262(15):7151-6. PMID 3584110
- [Background] Stewart AF, Wu T, Goumas D, Burtis WJ, Broadus AE. N-terminal amino acid sequence of two novel tumor-derived adenylate cyclase-stimulating proteins: identification of parathyroid hormone-like and parathyroid hormone-unlike domains. Biochem Biophys Res Commun. 1987 Jul 31;146(2):672-8. doi: 10.1016/0006-291x(87)90581-x. PMID 3619898
- [Background] Wu TL, Vasavada RC, Yang K, Massfelder T, Ganz M, Abbas SK, Care AD, Stewart AF. Structural and physiologic characterization of the mid-region secretory species of parathyroid hormone-related protein. J Biol Chem. 1996 Oct 4;271(40):24371-81. doi: 10.1074/jbc.271.40.24371. PMID 8798692
- [Background] Cosman F, Shen V, Xie F, Seibel M, Ratcliffe A, Lindsay R. Estrogen protection against bone resorbing effects of parathyroid hormone infusion. Assessment by use of biochemical markers. Ann Intern Med. 1993 Mar 1;118(5):337-43. doi: 10.7326/0003-4819-118-5-199303010-00003. PMID 8430979
- [Background] Hodsman AB, Fraher LJ, Ostbye T, Adachi JD, Steer BM. An evaluation of several biochemical markers for bone formation and resorption in a protocol utilizing cyclical parathyroid hormone and calcitonin therapy for osteoporosis. J Clin Invest. 1993 Mar;91(3):1138-48. doi: 10.1172/JCI116273. PMID 8450043
- [Derived] Horwitz MJ, Tedesco MB, Sereika SM, Prebehala L, Gundberg CM, Hollis BW, Bisello A, Garcia-Ocana A, Carneiro RM, Stewart AF. A 7-day continuous infusion of PTH or PTHrP suppresses bone formation and uncouples bone turnover. J Bone Miner Res. 2011 Sep;26(9):2287-97. doi: 10.1002/jbmr.415. PMID 21544866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Starting in October 2006, 19 Healthy caucasian males & females between 24 - 35 yrs were screened. By November 2007 11 subjects were randomized and 10 completed the one week infusion study which was done on the Clinical and Translational Research Clinic (CTRC) at the University of Pittsburgh Medical Center (UPMC).
Pre-assignment Details: Candidates were non-smokers and females had negative pregnancy tests. Those on chronic medications with the exception of oral contraceptives or stable thyroid hormone replacement were excluded. Body mass index had to be less than 30, and all had normal screening labs.
Groups:
- Group 1: PTH (1-34) 2 picomoles (pmols)/kg/hr
- Group 2: PTH (1-34) 4 picomoles (pmols)/kg/hr
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eleven subjects received parathyroid hormone (1-34) infusions intravenously for one week.
Groups:
- Parathyroid Hormone - 2 Picomoles/kg/hr.: Subjects initially entering the study receive study drug Parathyroid Hormone (1-34) in intravenous doses beginning at 2 picomoles/kg/hr. Doses will be slowly and safely escalated in groups of 3 subjects.
- Parathyroid Hormone(1-34) - 4 Picomoles/kg/hr: Subjects received Parathyroid Hormone (1-34)intravenously at 4 picomoles/kg/hr.
- Total: Total of all reporting groups
Arm/Group | Parathyroid Hormone - 2 Picomoles/kg/hr. | Parathyroid Hormone(1-34) - 4 Picomoles/kg/hr | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicity
Description: DLT was defined as achieving one major criterion or two minor criteria rated at ≥ 2 on a scale of 0-5. The major criteria were defined as symptomatic orthostatic hypotension (systolic BP fall >30 mm/hg), tachycardia (pulse > 120), hypertension (systolic BP >160 mm/hg on 2 occasions), hypercalcemia (serum calcium ≥ 12 mg/dl), and hypophosphatemia (serum phosphorous < 1.5 mg/dl). Minor criteria included symptoms such as flushing, nausea, abdominal or muscle cramps, dizziness, lightheadedness, palpitations, etc.
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days
Measure: Number; unit: participants
Groups:
- Group 1: PTH(1-34) 2 picomols (pmols)/kg/hr
- Group 2: PTH(1-34) 4 picomoles/kg/hr for one week
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
participants | 0 | 2

2. Primary Outcome: Total Serum Calcium
Description: mg/dl
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
mg/dl
  Baseline | 9.33 (0.20) | 9.11 (0.16)
  11P Day 1 | 9.56 (0.19) | 9.78 (0.21)
  7 A Day 2 | 9.74 (0.15) | 10.06 (0.22)
  3P Day 2 | 10.14 (0.18) | 10.30 (0.26)
  11P Day 2 | 9.84 (0.15) | 10.38 (0.37)
  7A Day 3 | 10.10 (0.17) | 10.52 (0.34)
  3P Day 3 | 10.32 (0.26) | 10.66 (0.42)
  11P Day 3 | 9.72 (0.31) | 9.94 (0.26)
  7A Day 4 | 10.04 (0.33) | 9.88 (0.17)
  3P Day 4 | 9.94 (0.30) | 9.94 (0.23)
  11P Day 4 | 9.54 (0.29) | 9.56 (0.19)
  7A Day 5 | 10.16 (0.47) | 9.64 (0.28)
  3P Day 5 | 10.26 (0.38) | 9.72 (0.31)
  11P Day 5 | 9.82 (0.37) | 9.46 (0.23)
  7A Day 6 | 10.18 (0.33) | 9.92 (0.23)
  3P Day 6 | 10.28 (0.40) | 10.28 (0.19)
  11P Day 6 | 9.56 (0.37) | 9.60 (0.31)
  7A Day 7 | 10.18 (0.35) | 9.90 (0.17)
  3P Day 7 | 10.02 (0.39) | 9.98 (0.19)
  11P Day 7 | 9.82 (0.33) | 10.03 (0.18)
  7A Day 8 | 10.38 (0.31) | 10.50 (0.22)
  FOLLOW-UP | 9.50 (0.20) | 9.50 (0.12)
Statistical Analysis 1: Comparison: Group 1; Test type: Non-Inferiority or Equivalence — The study was designed as a standard dose-escalation study, dose-finding pilot study. The primary outcome measures were safety (hypercalcemia, hypophosphatemia and symptoms/hemodynamic measurements). A modified Fibronacci dose-escalation scheme was employed; p < .0001, Mixed Models Analysis — The reported p-value corresponds to the increase over time for the PTH 2 pmol group; The level of statistical significance was set at .05 (two-tailed)

3. Primary Outcome: Ionized Serum Calcium
Description: mg/dl
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
mg/dl
  Baseline | 4.72 (0.10) | 4.52 (0.05)
  11P Day 1 | 4.93 (0.14) | 4.54 (0.18)
  7 A Day 2 | 5.17 (0.09) | 5.04 (0.11)
  3P Day 2 | 5.08 (0.06) | 5.01 (0.12)
  11P Day 2 | 5.01 (0.15) | 4.97 (0.17)
  7A Day 3 | 5.21 (0.19) | 5.22 (0.19)
  3P Day 3 | 5.08 (0.09) | 5.11 (0.20)
  11P Day 3 | 4.80 (0.17) | 4.82 (0.07)
  7A Day 4 | 5.10 (0.09) | 4.90 (0.08)
  3P Day 4 | 4.86 (0.17) | 4.77 (0.09)
  11P Day 4 | 4.93 (0.15) | 4.70 (0.06)
  7A Day 5 | 5.18 (0.24) | 4.84 (0.05)
  3P Day 5 | 5.03 (0.18) | 4.91 (0.18)
  11P Day 5 | 4.90 (0.16) | 4.68 (0.11)
  7A Day 6 | 5.29 (0.20) | 4.95 (0.13)
  3P Day 6 | 5.17 (0.13) | 4.89 (0.08)
  11P Day 6 | 5.02 (0.18) | 4.82 (0.14)
  7A Day 7 | 5.20 (0.14) | 4.99 (0.19)
  3P Day 7 | 4.89 (0.12) | 4.88 (0.18)
  11P Day 7 | 5.15 (0.19) | 4.86 (0.14)
  7A Day 8 | 5.34 (0.18) | 5.28 (0.16)
  FOLLOW-UP | 4.79 (0.05) | 4.70 (0.12)
Statistical Analysis 1: Comparison: Group 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .0001, Mixed Models Analysis — The reported p-value corresponds to the increase over time for the PTH 2 pmol group; The level of statistical significance was set at .05 (two-tailed)

4. Primary Outcome: Serum Phosphorous
Description: mg/dl
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
mg/dl
  Baseline | 3.51 (0.30) | 3.45 (0.28)
  11P Day 1 | 4.16 (0.12) | 3.78 (0.19)
  7 A Day 2 | 3.78 (0.15) | 3.68 (0.16)
  3P Day 2 | 3.82 (0.15) | 3.44 (0.24)
  11P Day 2 | 3.86 (0.12) | 3.78 (0.11)
  7A Day 3 | 3.68 (0.16) | 3.58 (0.15)
  3P Day 3 | 3.68 (0.18) | 3.28 (0.12)
  11P Day 3 | 3.86 (0.09) | 3.60 (0.23)
  7A Day 4 | 3.58 (0.17) | 3.64 (0.18)
  3P Day 4 | 3.38 (0.16) | 3.22 (0.16)
  11P Day 4 | 3.76 (0.07) | 3.52 (0.24)
  7A Day 5 | 3.56 (0.14) | 3.72 (0.23)
  3P Day 5 | 3.70 (0.20) | 3.22 (0.24)
  11P Day 5 | 3.56 (0.10) | 3.64 (0.21)
  7A Day 6 | 3.86 (0.12) | 3.60 (0.09)
  3P Day 6 | 3.78 (0.21) | 3.03 (0.23)
  11P Day 6 | 3.70 (0.16) | 3.63 (0.09)
  7A Day 7 | 3.70 (0.22) | 3.90 (0.18)
  3P Day 7 | 3.12 (0.17) | 3.18 (0.11)
  11P Day 7 | 3.48 (0.11) | 3.55 (0.21)
  7A Day 8 | 3.82 (0.19) | 3.80 (0.09)
  FOLLOW-UP | 4.12 (0.18) | 3.64 (0.28)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Mixed Models Analysis — The reported p-value corresponds to change over time for the PTH 2 and PTH 4 pmol groups; The level of statistical significance was set at .05 (two-tailed)

5. Secondary Outcome: 1,25 Vitamin D
Description: pg/ml
Time Frame: baseline, daily up to Day 8 and follow-up
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
pg/ml
  baseline | 37.78 (4.71) | 39.18 (5.82)
  Day 2 | 40.90 (2.78) | 42.72 (7.60)
  Day 3 | 35.68 (2.94) | 41.74 (6.39)
  Day 4 | 27.70 (7.57) | 34.72 (6.91)
  Day 5 | 36.16 (2.38) | 31.53 (4.78)
  Day 6 | 38.00 (3.13) | 35.68 (3.39)
  Day 7 | 32.18 (3.41) | 28.48 (2.82)
  Day 8 | 34.78 (3.57) | 33.13 (3.56)
  follow-up | 37.06 (4.46) | 40.16 (4.46)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .01, Mixed Models Analysis — The reported p-value corresponds to change over time for the PTH 2 and PTH 4 pmol groups; The level of statistical significance was set at .05 (two-tailed)

6. Secondary Outcome: Parathyroid Hormone (1-84)
Description: pg/ml
Time Frame: baseline, daily up to Day 8 and follow-up
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
pg/ml
  baseline | 20.90 (3.85) | 52.44 (12.88)
  Day 2 | 3.86 (0.86) | 5.30 (2.11)
  Day 3 | 3.00 (0.00) | 3.38 (0.38)
  Day 4 | 4.12 (1.12) | 5.00 (2.00)
  Day 5 | 4.64 (1.64) | 11.68 (6.28)
  Day 6 | 3.50 (0.50) | 6.34 (3.73)
  Day 7 | 3.58 (0.58) | 6.68 (3.68)
  Day 8 | 3.09 (0.09) | 3.00 (0.00)
  follow-up | 23.60 (2.29) | 35.20 (3.79)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .05, Mixed Models Analysis — the reported p-values correspond to the decrease compared to baseline in all arms/groups at Days 2-8; The level of statistical significance was set at .05 (two-tailed)

7. Secondary Outcome: Fractional Excretion of Calcium
Description: % = (S Creatinine X U Calcium)/(S Calcium X U Creatinine)
Time Frame: baseline and daily
Measure: Mean (Standard Error); unit: % of excretion
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
% of excretion
  baseline | 3.38 (1.42) | 1.80 (0.41)
  Day 2 | 2.83 (0.27) | 2.87 (0.71)
  Day 3 | 4.28 (0.63) | 3.76 (0.63)
  Day 4 | 2.82 (0.51) | 3.87 (0.89)
  Day 5 | 3.90 (0.69) | 2.54 (0.42)
  Day 6 | 4.44 (0.57) | 3.49 (0.69)
  Day 8 | 5.54 (0.70) | 4.58 (0.96)
Statistical Analysis 1: Comparison: Group 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .002, Mixed Models Analysis — the reported p-value corresponds to the increase compared to baseline over time (days 2-8) in the PTH 2 pmol group; The level of statistical significance was set at .05 (two-tailed)

8. Secondary Outcome: 24 Hour Urine Calcium
Description: mg/gm creatinine
Time Frame: 24 hours period from Day 7 to Day 8
Measure: Mean (Standard Error); unit: mg/gm creatinine
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
mg/gm creatinine | 315.278845 (25.0352949) | 210.24827 (58.3459645)

9. Secondary Outcome: Tubular Maximum for Phosphorous
Description: mg/dl
Time Frame: baseline and daily
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
mg/dl
  baseline | 3.80 (0.40) | 3.50 (0.28)
  Day 2 | 3.28 (0.16) | 3.30 (0.13)
  Day 3 | 3.37 (0.20) | 3.11 (0.24)
  Day 4 | 3.25 (0.27) | 3.66 (0.37)
  Day 5 | 3.19 (0.20) | 3.31 (0.22)
  Day 6 | 3.45 (0.16) | 3.25 (0.17)
  Day 8 | 3.52 (0.34) | 3.43 (0.10)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .61, Mixed Models Analysis — The reported p-value corresponds to change over time for the PTH 2 and PTH 4 pmol groups; The level of statistical significance was set at .05 (two-tailed)

10. Secondary Outcome: Serum Amino-terminal of Collagen- (sNTX)
Description: % change from baseline
Time Frame: baseline, daily, one week follow-up
Measure: Mean (Standard Error); unit: % change from baseline
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
% change from baseline
  baseline | 0 (0) | 0 (0)
  Day 2 | 61.8428952 (18.6263576) | 77.4709521 (13.5088219)
  Day 3 | 85.7699521 (27.761763) | 85.9288044 (12.9913176)
  Day 4 | 96.3668762 (29.0312368) | 59.9595445 (18.6508014)
  Day 5 | 107.517148 (29.2958519) | 83.3701575 (21.9993233)
  Day 6 | 150.594712 (38.2863053) | 120.268081 (17.8645936)
  Day 7 | 141.193285 (28.7484727) | 109.660098 (30.4136118)
  Day 8 | 153.72039 (38.1279427) | 148.451289 (23.0512356)
  follow-up | 4.06445076 (8.25178671) | 1.05486408 (11.8266679)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .008, Mixed Models Analysis — The reported p-value corresponds to the % increase compared to baseline in all Arms/groups on Days 2-8; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Mixed Models Analysis — The reported p-value corresponds the the % change from baseline at follow-up in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

11. Secondary Outcome: Serum Carboxy-terminal of Collagen- 1(sCTX)
Description: % change from baseline
Time Frame: baseline, daily, one week follow-up
Measure: Mean (Standard Error); unit: % change from baseline
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
% change from baseline
  baseline | 0 (0) | 0 (0)
  Day 2 | 113.70 (37.63) | 104.07 (11.83)
  Day 3 | 136.76 (45.34) | 112.11 (22.41)
  Day 4 | 142.66 (46.55) | 70.74 (37.02)
  Day 5 | 165.97 (55.34) | 92.13 (36.22)
  Day 6 | 205.39 (60.11) | 141.66 (17.80)
  Day 7 | 206.06 (60.02) | 168.77 (31.35)
  Day 8 | 225.04 (63.07) | 244.50 (25.28)
  follow-up | -6.78 (13.40) | -11.82 (17.86)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .0001, Mixed Models Analysis — The reported p-value corresponds to % change (increase) from baseline in all Arms/groups at Days 2-8; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Mixed Models Analysis — The reported p-value corresponds the the % change from baseline at follow-up in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

12. Secondary Outcome: Amino-terminal Peptides of Procollagen- 1(P1NP)
Description: % change from baseline
Time Frame: baseline, daily, one week follow-up
Measure: Mean (Standard Error); unit: % change from baseline
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
% change from baseline
  baseline | 0 (0) | 0 (0)
  Day 2 | -18.536953 (3.06129512) | -16.118573 (9.23396676)
  Day 3 | -31.14427 (3.986728) | -35.577655 (3.47737847)
  Day 4 | -32.942391 (1.15253446) | -35.018736 (5.91933273)
  Day 5 | -31.506308 (2.94297475) | -35.309609 (6.61031904)
  Day 6 | -36.35864 (5.71685066) | -35.064188 (5.84391487)
  Day 7 | -40.709396 (5.7024817) | -30.58629 (3.41615735)
  Day 8 | -39.046467 (4.79183284) | -35.619862 (3.18918608)
  follow-up | 31.4333667 (9.87895156) | 26.3367446 (16.1801142)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .0001, Mixed Models Analysis — the reported p-value corresponds to % decrease compared to baseline at Days 2-8 in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .01, Mixed Models Analysis — the reported p-value corresponds to % change from baseline at the follow-up visit in all Arms/groups; the reported p-value corresponds to % change from baseline at the follow-up visit in all Arms/groups

13. Secondary Outcome: Bone Specific Alkaline Phosphatase (BSAP)
Description: % change from baseline
Time Frame: baseline, daily, one week follow-up
Measure: Mean (Standard Error); unit: % change from baseline
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 5
% change from baseline
  baseline | 0 (0) | 0 (0)
  Day 2 | 7.35 (3.22) | 7.91 (7.47)
  Day 3 | -5.61 (4.67) | 9.05 (12.82)
  Day 4 | 4.34 (4.85) | 0.77 (9.93)
  Day 5 | -8.75 (3.39) | -2.19 (14.10)
  Day 6 | -3.42 (15.55) | -8.89 (11.60)
  Day 7 | -1.35 (12.69) | -13.72 (12.96)
  Day 8 | 2.09 (11.94) | -9.91 (16.98)
  follow-up | 14.08 (9.96) | 5.51 (8.28)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > .05, Mixed Models Analysis — the reported p-value corresponds to % change compared to baseline at Days 2-8 in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

ADVERSE EVENTS:
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=6) | Group 2 (N=5)
hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1)
tachycardia (Endocrine disorders) | 0 (0) | 1 (1)
IV infiltration (Endocrine disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small number of subjects in each group Study limited to Caucasians Only one timepoint for follow-up was measure Study did not include saline infused controls

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No